CLINICAL TRIAL: NCT06416800
Title: An Open-Label Study to Assess the Effect of Povorcitinib on Digoxin, Rosuvastatin, and Metformin Pharmacokinetics and the Effect of Probenecid on Povorcitinib Pharmacokinetics When Administered Orally to Healthy Adult Participants
Brief Title: A Study to Assess the Effect of Povorcitinib on Digoxin, Rosuvastatin, and Metformin Pharmacokinetics and the Effect of Probenecid on Povorcitinib Pharmacokinetics When Administered Orally to Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB54707-110
Record Dates: First submitted 2024-04-29; First posted 2024-05-16 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants
Keywords: INCB054707
MeSH Terms: interventions — Digoxin; Rosuvastatin Calcium; Metformin; Probenecid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Dose (Experimental): Digoxin and povorcitinib will be administered at protocol defined doses.
  Interventions: Drug: Digoxin; Drug: Povorcitinib
- Cohort 2: Dose (Experimental): Rosuvastatin and povorcitinib will be administered at protocol defined doses.
  Interventions: Drug: Rosuvastatin; Drug: Povorcitinib
- Cohort 3: Dose (Experimental): Metformin and povorcitinib will be administered at protocol defined doses.
  Interventions: Drug: Metformin; Drug: Povorcitinib
- Cohort 4: Dose (Experimental): Probenecid and povorcitinib will be administered at protocol defined doses.
  Interventions: Drug: Povorcitinib; Drug: Probenecid

INTERVENTIONS:
Drug: Digoxin — Oral; Tablet
  Arms: Cohort 1: Dose
Drug: Rosuvastatin — Oral; Tablet
  Arms: Cohort 2: Dose
Drug: Metformin — Oral; Tablet
  Arms: Cohort 3: Dose
Drug: Povorcitinib — Oral; Tablet
Drug: Probenecid — Oral; Tablet
  Arms: Cohort 4: Dose

SUMMARY:
The purpose of this study is to Assess the Effect of Povorcitinib on Digoxin, Rosuvastatin, and Metformin Pharmacokinetics and the Effect of Probenecid on Povorcitinib Pharmacokinetics When Administered Orally to Healthy Adult Participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Aged 18 to 55 years, inclusive, at the time of signing the ICF.
* BMI between 18.0 and 30.5 kg/m2, inclusive. Participants with a BMI up to 32.0 kg/m2 may be enrolled with the sponsor's approval.
* No clinically significant findings on screening evaluations (eg, clinical, laboratory, and ECG evaluations).
* Ability to swallow and retain oral medication.
* Willingness to avoid pregnancy or fathering children based on the criteria below:

  * Male participants with reproductive potential must agree to take appropriate precautions to avoid fathering children from screening through 90 days (a spermatogenesis cycle) after the last dose of study treatment and must refrain from donating sperm during this period. Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Female participants must have a negative serum pregnancy test at screening and a negative urine pregnancy test at check-in on Day -1 and must agree to take appropriate precautions to avoid pregnancy from screening through 30 days (1 menstrual cycle) after the last dose of study treatment and must refrain from donating oocytes during this period. Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Female participants not considered to be of childbearing potential are eligible.

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening.
* History of cardiovascular, cerebrovascular, peripheral vascular, or thrombotic disease or uncontrolled hypertension (ie, systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg at screening, confirmed by repeat testing).
* History or presence of cardiovascular symptoms including but not limited to chest pain or pressure, palpitations, irregular heartbeat, syncope (excluding vasovagal from phlebotomy), dyspnea at rest or on exertion, lightheadedness, orthopnea, or paroxysmal nocturnal dyspnea that is considered clinically significant by the investigator.
* Resting pulse < 40 bpm or > 100 bpm at screening, confirmed by repeat testing.
* History or presence of an abnormal ECG before initial dose administration that, in the investigator's opinion, is clinically significant (ie, a QTcF interval > 450 milliseconds for males and > 470 milliseconds for females, QRS interval > 120 milliseconds, and PR interval > 220 milliseconds).
* Presence or history of a malabsorption syndrome (eg, Crohn's disease or chronic pancreatitis) that could affect drug absorption.
* Hemoglobin, WBC count, platelet count, or absolute neutrophil count less than the laboratory LLN at screening or check-in, confirmed by repeat testing. Hemoglobin, WBC, platelet, and neutrophil abnormalities must also be clinically significant in the opinion of the investigator to be exclusionary.
* Vitamin B12, folate, TSH, or parathyroid hormone levels less than the laboratory LLN at screening that are also clinically significant in the opinion of the investigator.
* ALT, AST, ALP, or total bilirubin > 1.25 × the laboratory-defined ULN at screening or check-in, confirmed by repeat testing (except participants with Gilbert's disease, for whom total bilirubin must be ≤ 2.0 × ULN).
* History of malignancy within 5 years before screening, with the exception of cured basal cell or squamous cell carcinoma of the skin, ductal carcinoma in situ, or Gleason 6 prostate cancer.
* Current or recent (within 3 months before screening) clinically significant gastrointestinal disease or surgery (including cholecystectomy; excluding appendectomy) that could affect drug absorption.
* Any major surgery within 4 weeks of screening.
* Donation of blood to a blood bank or participation in a clinical study (except a screening visit) within 4 weeks before screening (within 2 weeks for plasma-only donation).
* Blood transfusion within 4 months before check-in (Day -1).
* Chronic or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment (includes latent treated tuberculosis).
* Positive test for HBV, HCV, or HIV. Participants whose results are compatible with prior immunization for or immunity due to infection with HBV may be included at the discretion of the investigator.
* Receipt of live (including attenuated) vaccines within 28 days before the first dose of study treatment or anticipation of need for such a vaccine during the study. Note: Nonlive or inactivated vaccines are allowed up to 2 weeks before the first dose of study treatment.
* History of significant alcohol use within 3 months before screening.
* Positive urine or breath test for ethanol or positive urine or serum screen for drugs of abuse that are not otherwise explained by permitted concomitant medications or diet.
* Current treatment, or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study treatment, with another investigational medication or current enrollment in another investigational drug study.
* Current treatment, or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study treatment, with an inducer or inhibitor of CYP3A4, P-gp, or BCRP (refer to the Drug Interaction Database [2024] for prohibited drugs).
* Consumption of Seville oranges, grapefruit or grapefruit juice, pomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices within 72 hours before the first dose of study treatment.
* Current use of prohibited medication.
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) deemed clinically relevant by the investigator.
* Known hypersensitivity or severe reaction to povorcitinib or any excipients of povorcitinib, digoxin, rosuvastatin, metformin or probenecid (refer to the IB and applicable package inserts).
* Inability to undergo venipuncture or tolerate venous access.
* History of tobacco- or nicotine-containing product-use within 1 month before screening. However, use of nicotine-containing products prior to screening that is equivalent to ≤ 2 cigarettes per week may be permitted at the discretion of the investigator.
* Use of prescription drugs (including hormonal contraceptives) within 14 days before study treatment administration or nonprescription medications/products (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days of study treatment administration. However, occasional paracetamol, ibuprofen, and standard-dose multivitamins are permitted.
* Women who are pregnant or breastfeeding.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study treatment and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* An eGFR < 90 mL/min/1.73 m2, based on the site's standard formula, at screening. A repeat measurement may be allowed at the investigator's discretion.
* Cohort 4 only: Uric acid levels less than the laboratory LLN at screening or check-in, confirmed by repeat testing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) in plasma digoxin | Up to Day 15
  Digoxin concentration in plasma.
PK in plasma rosuvastatin | Up to Day 11
  Rosuvastatin concentration in plasma.
PK in plasma metformin | Up to Day 14
  Metformin concentration in plasma.
PK in plasma povorcitinib | Up to Day 17
  Povorcitinib concentration in plasma.

SECONDARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to Day 25 (Cohorts 1, 3 and 4), Up to Day 22 (Cohort 2)
  Defined as any adverse event, either reported for the first time or the worsening of a pre-existing event, occurring after first dose of study treatment.
Additional digoxin PK parameters in plasma | Up to Day 15
  Additional digoxin concentration in plasma.
Additional rosuvastatin PK parameters in plasma | Up to Day 11
  Additional rosuvastatin concentration in plasma.
Additional metformin PK parameters in plasma | Up to Day 14
  Additional metformin concentration in plasma.
PK in plasma povorcitinib | Up to Day 15
  Povorcitinib concentration in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (1):
- Fortrea Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Assess the Effect of Povorcitinib on Digoxin, Rosuvastatin, and Metformin Pharmacokinetics and the Effect of Probenecid on Povorcitinib Pharmacokinetics When Administered Orally to Healthy Adult Participants — https://www.incyteclinicaltrials.com/study/?id=INCB54707-110&SearchTerm=INCB54707-110&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=